CLINICAL TRIAL: NCT00359515
Title: Mutation Detection for Lowe Syndrome
Brief Title: Genetic Analysis of Oculocerebrorenal Syndrome of Lowe
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010095; 01-HG-0095
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-03

CONDITIONS: Lowe Syndrome
Keywords: Archived Samples; Mutation Screening; Genotype-Phenotype Correlation; Pediatric Developmental Disorder; Cataracts; Mutation Detection; Lowe Syndrome; Genotype
MeSH Terms: conditions — Oculocerebrorenal Syndrome; Cataract

SUMMARY:
This study will investigate the genetic basis of oculocerebrorenal syndrome of Lowe (OCRL)-a rare X-linked disorder (carried by females and passed to males). Patients with OCRL have abnormal development of the eye lens, developmental delay, muscle weakness and kidney dysfunction.

The study will examine DNA and cell samples obtained and archived from patients with OCRL enrolled in a previous protocol (HG008A) between 1996 and 1999. It will identify mutations in the OCRL1 gene responsible for OCRL in affected males and try to correlate them with specific biochemical or cellular activities (e.g., enzyme activity, protein stability, cellular localization and trafficking). When test results are available, the information will be communicated to the patients, their parents (if the patient is a minor) and their physicians, and families will receive genetic counseling.

DETAILED DESCRIPTION:
Oculocerebrorenal syndrome of Lowe (OCRL) is a rare X-linked disorder characterized by congenital cataracts, mental retardation, and renal tubular dysfunction. Patients with known or suspected OCRL were enrolled under previous protocol 96-HG-0008 that expired in 1998 and was not renewed. We are continuing studies of DNA and cell samples obtained and archived under our previous protocol to identify mutations in the OCRL1 gene responsible for Lowe syndrome and related disorders in affected males and attempt to correlate these mutations to particular biochemical or cellular phenotypes (enzyme activity, protein stability, cellular localization and trafficking). Information about genotypes will not be communicated back to the patients, their parents (if patient is a minor) or their physicians as part of this study.

We are also continuing our investigations of heterogeneity in OCRL by studying collected cell cultures from our collaborator Dr. Steven Scheinman at Suny New York Medical University, Syracuse, from a group of patients with mutations in OCRL1 who have Dent disease, characterized by renal tubular dysfunction. These data, and the variability in the renal and CNS abnormalities that occur in OCRL are evidence for the existence of modifiers. We propose to identify genes that are differentially expressed in cells from OCRL patients, patients with Dent disease and OCRL1 mutations by gene expression analysis of RNA from patient samples.

As part of our study on phenotypic and genetic heterogeneity in OCRL, mutation analysis resulted in the identification of mutations mostly in the second two-thirds of OCRL1. However, the OCRL1 mutations in the Dent disease patients have been found in the first third of OCRL1. We plan to send samples from Lowe syndrome patients without identified OCRL1 mutations to a Dr. Steven Scheinman who will look for such OCRL1 mutations. He will be sent only coded samples and will look for such OCRL1 mutations. He will be sent only coded samples and will not have access to patient identifiers. This information will be used for research purposes only.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male gender, history of congenital cataracts, proximal renal tubular dysfunction, and developmental delay.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2001-02-17; Study Completion 2009-02-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States